CLINICAL TRIAL: NCT03361722
Title: Interest of Tissue Oxygen Pressure (PtiO2) Monitoring to Detect a Vasospasm Post Aneurysmal Subarachnoid Hemorrhage
Acronym: O2-VASO
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: CE_20151215_1_SWG
Record Dates: First submitted 2017-11-29; First posted 2017-12-05 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-11

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Vasospasm is a current complication after aneurysmal subarachnoid hemorrhage and often and often associated with brain ischemia. This complication is difficult to detect, because clinical examination is hardly helpful in sedated patients and the performances of transcranial doppler can only detect the spasm of middle cerebral arteries.

Tissue Oxygen Pressure (PtiO2) Monitoring allows early detection of brain oxygenation local modifications and of brain ischemia, via continuous monitoring.

This study aims to assess the performance of the tissue oxygen pressure monitoring in detecting a vasospasm post aneurysmal subarachnoid hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* severe aneurysmal subarachnoid hemorrhage
* patient sedated
* patient hospitalized in intensive care unit between January 2013 and August 2015
* multimodal neurologic monitoring including Tissue Oxygen Pressure and transcranial doppler

Exclusion Criteria:

* insonation impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients, hospitalized in intensive care unit and sedated, with severe aneurysmal subarachnoid hemorrhage
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-02-15 (Actual); Primary Completion 2016-09-15 (Actual); Study Completion 2016-09-15 (Actual)

PRIMARY OUTCOMES:
Tissue Oxygen Pressure | baseline